CLINICAL TRIAL: NCT07118111
Title: The Role of Resin Infiltration Treatment on Dental Hypersensitivity and Patient-Parent Satisfaction in Children With Anterior Teeth Affected by Hypomineralization or Hypoplasia
Brief Title: Effect of Resin Infiltration on Hypersensitivity and Satisfaction in Children With Enamel Defects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gizem Tıraşçı (Other)
Responsible Party: Sponsor-Investigator, Gizem Tıraşçı, Research Assistant, Inonu University
Organization: Inonu University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/7696
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Molar Incisor Hypomineralisation; Enamel Hypoplasia; Dental Hypersensitivity
Keywords: resin infiltration; hypomineralization; hypoplasia; dental sensitivity
MeSH Terms: conditions — Molar Hypomineralization; Dental Enamel Hypoplasia

STUDY DESIGN:
Intervention Model Description: This is a single group interventional study where all participants receive resin infiltration treatment. There is no comparison or control group. Outcomes such as dental hypersensitivity and patient satisfaction will be measured before and after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resin Infiltration Treatment Group (Other): All participants receive resin infiltration treatment to anterior teeth affected by enamel defects.
  Interventions: Procedure: Resin infiltration

INTERVENTIONS:
Procedure: Resin infiltration — Application of a low-viscosity resin infiltrant to the anterior teeth affected by enamel defects. This procedure aims to reduce dental hypersensitivity and improve esthetic appearance.

SUMMARY:
This study evaluates the effect of resin infiltration on dental sensitivity, quality of life, and satisfaction in children aged 7-14 with enamel defects in their front teeth. Forty children received treatment, and outcomes were measured through sensitivity tests and questionnaires for both children and parents.

DETAILED DESCRIPTION:
Developmental enamel defects can negatively impact oral health-related quality of life by causing esthetic concerns and dental hypersensitivity in children. This prospective clinical study included 40 children aged 7-14 years diagnosed with hypomineralization or hypoplasia in their anterior teeth. All participants received resin infiltration treatment. Dental hypersensitivity was evaluated pre- and post-treatment using the Schiff Cold Air Sensitivity Scale (SCASS). Oral health-related quality of life was assessed using the Pediatric Oral Health-Related Quality of Life (POQL) scale through both child and parent forms. Post-treatment esthetic satisfaction levels were recorded based on reports from both children and their parents. The study aimed to determine the impact of resin infiltration on improving sensitivity, quality of life, and satisfaction in this population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 7 and 14 years.
* Children in good general health without any systemic disease.
* Presence of at least one anterior permanent tooth with hypomineralization or hypoplasia.
* Teeth with lesions larger than 1 mm that are suitable for resin infiltration treatment.
* Voluntary participation of both the child and their parent/guardian in the study, with signed informed consent.

Exclusion Criteria:

* Children with systemic diseases or undergoing medical treatment.
* Cases with active caries, trauma, restorations, or endodontic treatment applied or required on anterior teeth.
* Individuals who have previously received resin infiltration or similar treatment on the same tooth.
* Children with a history of allergies or sensitivity to the materials used in the procedure.
* Individuals who have received interventions such as fluoride varnish, fissure sealants, or tooth whitening on their teeth.
* Children who do not possess the cognitive ability to understand and respond to the questionnaire or sensitivity assessment.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Dental Hypersensitivity and Patient-Parent Satisfaction | Baseline, 1 month, 3 months, and 6 months after treatment
  Dental hypersensitivity will be assessed using the Schiff Cold Air Sensitivity Scale (SCASS) before treatment and at 1, 3, and 6 months post-treatment, where higher scores indicate greater sensitivity. Patient and parent satisfaction regarding esthetic and functional outcomes will be measured through standardized questionnaires administered after treatment.
  Schiff Cold Air Sensitivity Scale (SCASS):
  0 - The patient does not respond to the air stimulus.
  1. - The patient is aware of the stimulus but does not indicate discomfort and does not request discontinuation.
  2. - The patient responds to the stimulus with clear discomfort and requests discontinuation, either verbally or by turning the head.
  3. - The patient responds to the stimulus with pain and immediately and clearly requests discontinuation.
Change in Dental Hypersensitivity and Patient-Parent Satisfaction | 1 month, 3 months, and 6 months after treatment
  Dental hypersensitivity will be assessed using the Schiff Cold Air Sensitivity Scale (SCASS) before treatment and at 1, 3, and 6 months post-treatment, where higher scores indicate greater sensitivity. Patient and parent satisfaction regarding esthetic and functional outcomes will be measured through standardized questionnaires administered after treatment.
  Schiff Cold Air Sensitivity Scale (SCASS):
  0 - The patient does not respond to the air stimulus.
  1. - The patient is aware of the stimulus but does not indicate discomfort and does not request discontinuation.
  2. - The patient responds to the stimulus with clear discomfort and requests discontinuation, either verbally or by turning the head.
  3. - The patient responds to the stimulus with pain and immediately and clearly requests discontinuation.

SECONDARY OUTCOMES:
ral Health-Related Quality of Life, Esthetic Evaluation, Treatment Compliance | Baseline, 1 month, 3 months, and 6 months after treatment
  Oral health-related quality of life (OHRQoL) will be measured using the Pediatric Oral Health-Related Quality of Life (POQL) scale completed by both children and their parents before treatment and at follow-up visits. POQL scores will be calculated on a 0-100 scale, with higher scores indicating a lower quality of life. Esthetic changes will be assessed via clinical evaluations and patient/parent satisfaction surveys. Treatment compliance and acceptability will be recorded during the intervention process. Any adverse effects or complications following resin infiltration treatment will be monitored and documented throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sacide DUMAN, DDS, Study Director — Inonu University
Locations (1):
- Inonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to patient confidentiality concerns and restrictions imposed by the informed consent forms. Additionally, the data contain sensitive personal health information, and sharing is limited to protect participant privacy in accordance with ethical guidelines and institutional policies.